CLINICAL TRIAL: NCT00401063
Title: Acupuncture Case Series: Cancer Pain and Quality of Life
Brief Title: Usefulness of Acupuncture in Cancer Pain and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sivarama Vinjamury, Professor, Southern California University of Health Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCU-06-VINJ001
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Cancer; Pain
Keywords: Cancer; Acupuncture; Cancer Pain; Quality of life
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): Acupuncture treatment
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture treatment twice a day for eight weeks

SUMMARY:
The purpose of this study is to assess the effects of acupuncture on aspects of health including pain, energy level, sleep quality, activities of daily living and appetite.

DETAILED DESCRIPTION:
After receiving permission from the attending physician each study participant who meets the inclusion criteria will then undergo a physical examination and fill out several questionnaires. Each participant will undergo one to three treatments per week for a period of eight weeks. There will be one follow-up visit on the twelfth week. Participation in this study is free of charge, including all exams, treatment and informational material.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cancer by an MD/oncologist
* Age of 18 or older
* Baseline pain score of 3 or above on 0-10 rating scale
* In the evaluation of the treating physician or medically-qualified investigator, the patient's pain syndrome is the result of underlying cancer or cancer treatment
* Being ambulatory
* Permission from the treating physician (MD/oncologist)
* Platelet count of 50,000 or greater

Exclusion Criteria:

* Acupuncture treatment in past four weeks
* Neutropenia defined as ANC (absolute neutrophil count) < 1000/ml
* Inability to obtain permission from the treating physician
* Unwillingness to sign informed consent form
* Involvement in litigation
* Simultaneous infection with HIV or Hepatitis C virus
* Unable to present for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ-30 Quality of Life Questionnaire for Cancer Patients | Every two weeks, 0, 2, 4, 6, 8 and 12
Visual Analogue Scale | Every two weeks, 0,2,4,6,8, and 12 weeks

SECONDARY OUTCOMES:
BDI Psychological Assessment | Every two weeks, 0, 2, 4, 6, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sivarama P Vinjamury, MD, MAOM, Principal Investigator — Southern California University of Health Sciences
Locations (2):
- United States (2):
  - University Health Center, Pasadena, California
  - Southern California University of Health Sciences, Whittier, California

REFERENCES:
- See also: Visit Southern California University of Health Sciences Website — http://www.scuhs.edu